CLINICAL TRIAL: NCT05143632
Title: Continuous Non-invasive Blood Pressure Monitoring to Increase Hemodynamic Stability During Sitting Position Orthopedic Surgery: Prospective Randomized Study
Brief Title: Hemodynamic OptimizaTion in Sitting POsition Surgery Trial
Acronym: HOTSPOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, VERGARI ALESSANDRO, Aggregate Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HOTSPOT21
Record Dates: First submitted 2021-11-10; First posted 2021-12-03 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Hemodynamic Instability; Blood Pressure, Low; Orthopedic Disorder
MeSH Terms: conditions — Hypotension; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intermittent NIBP monitoring (No Intervention): Oscillometric intermittent (3 mins) noninvasive blood pressure monitoring
- ClearSight (Experimental): Continuous non invasive hemodynamic monitoring
  Interventions: Device: ClearSight

INTERVENTIONS:
Device: ClearSight — The primary hypothesis is that continuous non-invasive monitoring using ClearSight reduces the incidence of intraoperative hypotensive events (defined by mean arterial pressure below a value of 65 mmHg for more than 1 minute) and the duration of the events themselves, leading to an improvement in patients' outcomes.
  Arms: ClearSight

SUMMARY:
Intraoperative hypotension (MAP <65 mmHg) in patients undergoing general anesthesia is a notable risk factor for the development of post-operative complications including acute kidney injury (AKI), myocardial injury, stroke and delirium, and is strongly associated with increased mortality. Moreover, the mean and systolic blood pressure values tend to undergo significant fluctuations with different positions assumed by the patient during surgery. Since severe hypotensive phenomena are connected with cerebral hypoperfusion and are associated with negative outcomes, close monitoring of blood pressure is necessary.

The primary endpoint of this study is to evaluate the number of hypotensive episodes, their quality and their duration in patients monitored with the oscillometric intermittent noninvasive blood pressure method compared to patients with continuous noninvasive monitoring using ClearSight during orthopedic surgery in sitting position performed under general anesthesia and with interscalene block. The measure of hypotension will be expressed (in mmHg) with the TWA-MAP value (time-weighted average intraoperative MAP) to define the severity and duration of the hypotensive episode. Secondary endpoints include: episodes of cerebral desaturation measured by brain oximetry, number of severe hypotensive episodes (MAP <60 mmHg or <50 mmHg) recorded; time to event: how long does it take for the medical staff to correct the hypotensive episode (treated according to the planned protocol); quantity of vasopressors and/or fluids used to correct the hypotensive event; incidence of perioperative adverse cardiac events and acute kidney injury.

The primary hypothesis is that continuous non-invasive monitoring using ClearSight reduces the incidence of intraoperative hypotensive events (defined by mean arterial pressure below a value of 65 mmHg for more than 1 minute) and the duration of the events themselves, leading to an improvement in patients' outcomes.

DETAILED DESCRIPTION:
Intraoperative hypotension (MAP <65 mmHg) in patients undergoing general anesthesia is a notable risk factor for the development of post-operative complications including acute kidney injury (AKI), myocardial injury, stroke and delirium, and is strongly associated with increased mortality. Moreover, the mean and systolic blood pressure values tend to undergo significant fluctuations with different positions assumed by the patient during surgery, decreasing in the transition from the supine position to the sitting position (beach chair position) typically used during surgery that involves the anatomical district of the shoulder or proximal humerus. Since severe hypotensive phenomena are connected with cerebral hypoperfusion and are associated with negative outcomes, close monitoring of blood pressure is necessary. The investigators have introduced in clinical practice the use of non-invasive ClearSight sensor (Edwards Lifesciences Corp, Irvine CA, USA), which uses the volume-clamp and Physiocal technologies to obtain continuously calibrated blood pressure values and hemodynamic parameters. The primary endpoint of this study is to evaluate the number of hypotensive episodes, their quality and their duration in patients monitored with the oscillometric intermittent noninvasive blood pressure method compared to patients with continuous noninvasive monitoring using ClearSight during orthopedic surgery in seated position performed under general anesthesia and with interscalene block. The measure of hypotension will be expressed with the TWA-MAP value (time-weighted average intraoperative MAP) to define the severity and duration of the hypotensive episode. For a subgroup of patients, brain oximetry will be monitored using the ForeSight system to record episodes of cerebral desaturation. Secondary endpoints include: the incidence of brain oxygen desaturation measured using the ForeSight system, number of severe hypotensive episodes (MAP <60 mmHg or <50 mmHg) recorded; time to event: how long does it take for the medical staff to correct the hypotensive episode (treated according to the planned protocol); quantity of vasopressors and/or fluids used to correct the hypotensive event; incidence of perioperative adverse cardiac events and acute kidney injury.

The primary hypothesis is that continuous non-invasive monitoring using ClearSight reduces the incidence of intraoperative hypotensive events (defined by mean arterial pressure below a value of 65 mmHg for more than 1 minute) and the duration of the events themselves, leading to an improvement in patients' outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. patients candidate for elective orthopedic surgery in sitting position under general anesthesia + interscalene block

Exclusion Criteria:

1. non-elective patients (acute trauma) and hemodynamically unstable patients
2. vascular system pathologies
3. pregnant women
4. patient refusal to participate to the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
TWA MAP < 65 mmhg (expressed in mmHg) | Surgery time
  The measure of hypotension will be expressed with the TWA-MAP value (time-weighted average intraoperative MAP) in mmHg to define the severity and duration of the hypotensive episode. The TWA MAP under a threshold of 65 mmHg will be calculated as the area between 65 mmHg threshold and the curve of the MAP measurements divided by total continuous reading time in minutes.

SECONDARY OUTCOMES:
Incidence of cerebral oxygen desaturation episode | Surgery time
  The number of severe hypotensive episodes (StO2 <60%) recorded in the two groups.
Rate of severe hypotensive episodes (MAP <60 mmHg or <50 mmHg) | Surgery time
  The number of severe hypotensive episodes (MAP <60 mmHg or <50 mmHg) recorded.
Time to event (in seconds) | Surgery time
  How long does it take for the medical staff to correct the hypotensive episode (in seconds).

OTHER OUTCOMES:
Quantity of vasopressors and/or fluids | Surgery time
  Quantity of vasopressors (expressed in mg) and/or fluids (expressed in ml) used to correct the hypotensive events.
Incidence of perioperative adverse cardiac events. | 30 postoperative days.
  Major Adverse Cardiovascular Events - MACE - will be defined, according to the 3 points MACE, as a composite of non fatal stroke, non fatal myocardial infarction and cardiovascular death occurred within 30 postoperative days.
Incidence of perioperative acute kidney injury. | 48 postoperative hours.
  Acute Kidney Iniury - AKI - will be defined, according to the KDIGO criteria, as an increase in serum creatinine by greather than or equal to 0.3 mg/dL within 48 postoperative hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico A. Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vergari A, Frassanito L, Piersanti A, Vassalli F, Pitoni S, Ruggiero E, Nestorini R, Festa R, Bernardi G, Lombardo P, Caputo CT, Ciolli G, Rossi M. Continuous versus intermittent noninvasive blood pressure monitoring during beach chair position for shoulder surgery: A randomised controlled trial. Eur J Anaesthesiol. 2026 Feb 1;43(2):139-148. doi: 10.1097/EJA.0000000000002259. Epub 2025 Aug 22. PMID 40855940